CLINICAL TRIAL: NCT00031239
Title: Sleep Apnea in Look AHEAD Participants - Ancillary to Look AHEAD
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 994; R01HL070301 (NIH)
Record Dates: First submitted 2002-02-27; First posted 2002-02-28 (Estimated); Last update posted 2016-07-29 (Estimated); Status verified 2009-05

CONDITIONS: Sleep Apnea Syndromes; Diabetes Mellitus, Non-insulin Dependent; Obesity; Diabetes Mellitus
MeSH Terms: conditions — Sleep Apnea Syndromes; Diabetes Mellitus, Type 2; Obesity; Diabetes Mellitus

SUMMARY:
To assess the effects of weight loss on sleep disordered breathing in obese, Type 2 diabetics with obstructive sleep apnea.

DETAILED DESCRIPTION:
BACKGROUND:

Weight loss is a frequently recommended treatment for obese patients with obstructive sleep apnea (OSA). The empirical support for this recommendation is lacking. Based on descriptive studies, weight loss appears to improve but not abolish sleep disordered breathing. Moreover, the degree of improvement in OSA is quite variable and not directly proportional to weight loss. The lack of randomized trials, the study of predominantly male samples, and the absence of follow-up evaluations leave physicians and patients unsure about the utility of weight loss treatment in obese OSA patients.

The study is ancillary to the Look AHEAD clinical trial which is sponsored primarily by the National Institute of Diabetes and Digestive and Kidney Diseases and secondarily by the National Heart, Lung, and Blood Institute, the National Institute of Nursing Research, the Office of Research on Women's Health, the National Center on Minority Health and Health Disparities, and the Centers for Disease Control and Prevention. The Look AHEAD study is a multicenter, randomized clinical trial to examine the long-term effects of a lifestyle intervention designed to achieve and maintain weight loss in overweight diabetics.

DESIGN NARRATIVE:

The study will assess the effects of weight loss on sleep disordered breathing in 120 obese, Type 2 diabetics with obstructive sleep apnea (respiratory disturbance index [RDI] greater than or equal to 15) who are randomly assigned to either weight loss (n=60) or usual care (n=60) treatments within the context of the Look AHEAD study. Home polysomnography studies will be performed before treatment and at one and two years. Among the 60 weight loss subjects, the investigators will assess the relative importance of changes in neck and abdominal fat in explaining the variability of changes in sleep disordered breathing after weight loss. Finally, they will examine the relationship between changes in sleep-disordered breathing and changes in blood pressure after weight loss in the 60 weight loss participants. Specifically, this research will: 1) determine the efficacy of a weight loss program in reducing sleep disordered breathing in obese Type 2 diabetics; 2) identify sources of variability in sleep disordered breathing associated with weight loss; and 3) examine the role of sleep disordered breathing in mediating changes in blood pressure associated with weight loss. The results of this study will provide an empirical basis for making recommendations about the effectiveness of weight loss in Type 2 diabetics with OSA.

ELIGIBILITY:
An estimated 176 obese, diabetic subjects with obstructive sleep apnea, 50% women and 40% minorities.

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2001-09; Primary Completion 2006-07 (Actual); Study Completion 2006-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gary Foster — University of Pennsylvania

REFERENCES:
- [Background] Foster GD. Principles and practices in the management of obesity. Am J Respir Crit Care Med. 2003 Aug 1;168(3):274-80. doi: 10.1164/rccm.200205-456PP. No abstract available. PMID 12888610